CLINICAL TRIAL: NCT00506519
Title: Exploratory Efficacy and Safety, Pharmacokinetics and Dose Finding Study of ATryn® (Antithrombin Alfa) in Patients With Disseminated Intravascular Coagulation Associated With Severe Sepsis
Brief Title: Recombinant Human Antithrombin (ATryn®) in the Treatment of Patients With DIC Associated With Severe Sepsis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEO 90010-I21
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2021-08

CONDITIONS: Disseminated Intravascular Coagulation
Keywords: DIC associated with severe sepsis
MeSH Terms: conditions — Disseminated Intravascular Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AT-150 (Experimental): Loading dose followed by maintenance IV infusion for 5 days to maintain antithrombin activity at the target level 125-175%
  Interventions: Drug: Antithrombin alfa (INN name)
- AT-250 (Experimental): Loading dose followed by maintenance IV infusion for 5 days to maintain antithrombin activity at the target level 225-275%
  Interventions: Drug: Antithrombin alfa (INN name)
- Control (Active Comparator): The best standard treatment for the underlying condition only
  Interventions: Drug: Control (Standard treatment)

INTERVENTIONS:
Drug: Antithrombin alfa (INN name)
  Arms: AT-150; AT-250
Drug: Control (Standard treatment)
  Arms: Control

SUMMARY:
The primary objective of the study is to explore the efficacy and safety of ATryn® (antithrombin alfa) for the treatment of disseminated intravascular coagulation (DIC) associated with severe sepsis, when administered by continuous intravenous (IV) infusion over five days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent has been obtained from the patient or his/her legally acceptable representative
* Severe sepsis
* Disseminated intravascular coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AT-150: Loading dose followed by maintenance IV infusion for 5 days to maintain antithrombin activity at the target level 125-175%
  antithrombin alfa (INN name)
- AT-250: Loading dose followed by maintenance IV infusion for 5 days to maintain antithrombin activity at the target level 225-275%
  antithrombin alfa (INN name)
- Control: The best standard treatment for the underlying condition only
  Control
Period: Overall Study
Arm/Group | AT-150 | AT-250 | Control
Started | 10 | 10 | 5
Completed Treatment (Day 5) | 8 | 7 | 5
Day 28 Follow up | 8 | 6 | 5
Completed (Day 90 follow up (trial completed)) | 5 | 4 | 5
Not Completed | 5 | 6 | 0
Not completed — Death | 4 | 6 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AT-150 | AT-250 | Control | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (16.6) | 65.5 (19.4) | 58 (22.9) | 60.6 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 4 | 16
  Male | 2 | 6 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic origin: Caucasian | 8 | 10 | 5 | 23
  Ethnic origin: Asian | 2 | 0 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 75.6 (11.3) | 77.1 (14.5) | 71.4 (28.2) | 75.4 (16.2)
Height [Mean (Standard Deviation); unit: cm] | 163 (4.2) | 169 (14.1) | 161 (13.7) | 165 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Patients Alive on Day 28, Having Had an Improvement in the DIC Score (Overt or Non-overt) by at Least 2 Points Between Baseline and Day 6 and Having Had no Worsening of the SOFA Score Between Baseline and Day 6.
Description: Disseminated Intravascular Coagulation (DIC) ranges from 0 to 8 points, the higher the score the worse coagulation/outcome.
  Sepsis-related Organ Failure Assessment (SOFA) is a composite score of scores for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each system is scored from 0 to 4 with a higher score given for worse organ function. The scores are then added together to give a total range from 0 to 24 with a higher score representing a worse outcome.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Participants | 2 | 2 | 2

2. Secondary Outcome: Mortality at Day 28
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Participants | 1 | 4 | 0

3. Secondary Outcome: Mortality at Day 90
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Participants | 4 | 6 | 0

4. Secondary Outcome: Change From Baseline to Day 6 in SOFA Score Among Survivors on Day 6
Description: Sepsis-related Organ Failure Assessment (SOFA) is a composite score of scores for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each system is scored from 0 to 4 with a higher score given for worse organ function. The scores are then added together to give a total range from 0 to 24 with a higher score representing a worse outcome.
Time Frame: Baseline to Day 6
Population: Participants alive on day 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 9 | 7 | 5
score on a scale | -0.2 (1.2) | -0.3 (1.5) | 0.2 (1.1)

5. Secondary Outcome: Change From Baseline to Day 6 in DIC Score Among Survivors on Day 6
Description: Disseminated Intravascular Coagulation (DIC) ranges from 0 to 8 points, the higher the score the worse coagulation/outcome
Time Frame: Baseline to Day 6
Population: Participants alive on day 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 9 | 7 | 5
score on a scale | -3.0 (1.7) | -2.2 (2.4) | -3.0 (1.6)

6. Secondary Outcome: Days Alive and Out of ICU Day 28
Description: Days alive and out of ICU at day 28 for all patients
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Days | 9.8 (10.8) | 4.7 (10.0) | 13.6 (8.4)

7. Secondary Outcome: Days Alive and Out of Hospital Day 28
Description: Days alive and out of Hospital at day 28 for all patients
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Days | 3.0 (6.4) | 3.0 (6.6) | 4.6 (7.4)

8. Secondary Outcome: Days Alive and Free of Inotrope/Vasopressor Support Day 28
Description: Days alive and free of inotrope/vasopressor at day 28 for all patients
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Days | 20.7 (9.0) | 12.4 (11.7) | 21.6 (6.8)

9. Secondary Outcome: Days Alive and Off Ventilator Day 28
Description: Days alive and free of mechanical ventilation at day 28 for all patients
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Days | 11.4 (10.5) | 8.9 (11.8) | 14.4 (8.8)

10. Secondary Outcome: Days Alive and Free of Need for Renal Replacement Therapy Day 28
Description: Days alive and out of renal replacement therapy at day 28 for all patients
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Control: The best standard treatment for the underlying condition only
  Control (Standard treatment)
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 10 | 10 | 5
Days | 22.6 (13.3) | 10.5 (13.4) | 23.0 (6.9)

11. Secondary Outcome: Change From Baseline to Day 6 in Inflammation Marker IL-6
Time Frame: Baseline to Day 6
Population: Participants alive on day 6 who gave a sample.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 9 | 6 | 5
pg/mL | -68429 (192828) | -13153 (31801) | -69651 (141889)

12. Secondary Outcome: Change From Baseline to Day 6 in Inflammation Marker Procalcitonin
Time Frame: Baseline to Day 6
Population: Participants alive on day 6 who gave a sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AT-150 | AT-250 | Control
Number analyzed (Participants) | 9 | 6 | 5
ng/mL | -203.8 (340.2) | -51.1 (49.6) | -139.6 (146.2)

ADVERSE EVENTS:
Time Frame: 90 days
Description: In this study Critical events were defined to include major bleedings, thromboembolic complications and deaths and are reported as 'Serious Adverse Events'.
  All other adverse events were collected and reported together as 'Other (not including Serious) Adverse Events'.
Arm/Group | AT-150 | AT-250 | Control
All-Cause Mortality (participants affected / at risk) | 4/10 | 6/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/10 | 8/10 | 5/5
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT-150 (N=10) | AT-250 (N=10) | Control (N=5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 3 (8) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Tracheal haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Rectal haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (2)
Catheter site discharge (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 2 (2) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AT-150 (N=10) | AT-250 (N=10) | Control (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular bigeminy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Biloma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cytolytic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acquired hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Myocarditis septic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Blister (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Vitamin K decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalomyelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuromyopathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cortical necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site discharge (General disorders) | 0 (0) | 0 (0) | 1 (1)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Puncture site heamorrhage (General disorders) | 1 (1) | 0 (0) | 2 (2)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all clinical trials in peer-reviewed journals regardless of whether the findings are positive or negative, and acknowledges the investigators' right to publish results irrespective of outcome. Investigators are permitted to publish their individual data with the prior review and consent of LEO Pharma A/S